CLINICAL TRIAL: NCT06987500
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of XNW29016 Tablets in Advanced Solid Tumors With Failed Standard Treatment
Brief Title: A Study of PARG Inhibitor XNW29016 in Patients With Advanced Solid Tumors Who Failed Standard Treatment
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNW29016-I/II-01
Record Dates: First submitted 2025-04-25; First posted 2025-05-23 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase Ia: Monotherapy Dose Escalation (Experimental): Participants will receive XNW29016 at escalating dose levels
  Interventions: Drug: XNW29016
- Phase Ib: Monotherapy Dose Expansion (Experimental): The patient will be enrolled into several groups and take XNW29016 tablet twice a day. The subject of this part is to optimize dosage and definite RP2D.
  Interventions: Drug: XNW29016

INTERVENTIONS:
Drug: XNW29016 — Oral Medication. The study set 7 dose level cohorts in dose escalation part.
  Other Names: PARGi
  Arms: Phase Ia: Monotherapy Dose Escalation
Drug: XNW29016 — Oral Medication
  Other Names: PARGi
  Arms: Phase Ib: Monotherapy Dose Expansion

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, and efficacy of XNW29016 in participants with advanced solid tumors .

DETAILED DESCRIPTION:
This study is an open-label, multi-center Phase I/II clinical trial. Phase I includes the dose escalation (Stage Ia) and dose expansion (Stage Ib) phases; Phase II is an open-label, multi-center, single-arm basket study to evaluate the efficacy and safety of XNW29016 tablets in subjects with the target indications.

This study consists of a screening period, a treatment period, and a follow-up period. Subjects who meet the eligibility criteria during the screening period will enter the treatment period and receive treatment with XNW29016 tablets until the study treatment is discontinued due to reasons such as disease progression or intolerable toxicity.

Safety data (such as routine blood tests, routine biochemical tests, ECG, etc.) will be continuously collected during the study, and blood samples for PK (pharmacokinetics), PD (pharmacodynamics), etc. will also be collected. Efficacy evaluation will be based on different tumor types and collect different indicators. The efficacy evaluation will be conducted once every 8 weeks in the first 48 weeks from the start of the study treatment, and then once every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and sign an approved informed consent form (ICF).
* Age at the time of consent ≥ 18 years;
* Life expectancy of ≥ 3 months;
* For prostate adenocarcinoma, at least one evaluable lesion by RECIST v1.1 and PCWG3 criteria; for other advanced solid tumor, at least one measurable lesion by RECIST v1.1 criteria.
* Agree to provide tumor tissue samples that meet the testing requirements;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
* Phase Ia：Patients with advanced solid tumor confirmed by histological or cytological examination,who have failed standard of care therapy, or are unable to tolerate standard of care therapy, or unable to obtain/unwilling to receive standard therapy.
* Adequate hematologic and non-hematologic function during the screening.
* Women of childbearing potential must have a negative result of serum pregnancy test at screening, and must agree to use a reliable and effective method of contraception during the study and for 6 months after the last dose of the study drug. Male patients must agree to take adequate contraceptive measures from the beginning of the study to at least 6 months after the last dose of the test drug, and prohibit sperm donation;
* Ability to comply with all procedures of the clinical trial protocol.

Exclusion Criteria:

* Any previous treatment with a PARG inhibitor.
* Subjects known to be allergic to the study drug or its active ingredients or excipients;
* Subjects who received anti-tumor therapies including chemotherapy, immunotherapy, radical radiotherapy, major surgery, targeting therapy and other anti-tumor therapies within 4 weeks or 5 half-lives of the drug (whichever is shorter) before the first dose; or received palliative radiotherapy within 2 weeks before the first dose;
* Subjects who participated in any other clinical trial of anti-tumor therapy within 28 days before the first dosing, and the last dose of other anti-tumor trial drug is within 28 days prior to the first administration of study drug in this trial;
* Subjects who underwent major surgery within 4 weeks prior to the start of the study treatment, or who are scheduled to undergo a major surgery during the study period (procedures such as puncture or lymph node biopsy is allowed);
* Subjects who have an allogeneic tissue/ solid organ transplantation;
* Subjects who experienced toxicity events during previous anti-tumor treatment and the toxicity has not resolved (the toxicity events has not been graded as ≤ level 1 according to NCI-CTCAE 5.0). Other toxicities that the investigator does not think it will affect the safety assessment of the subject (such as hair loss, etc.) will be allowed;
* Subjects who have a history of other malignancies within 3 years prior to enrollment and do not meet the criteria for clinical cure.
* Central nervous system metastasis or disease;
* Subjects who have impaired heart functions or clinically serious heart disease；
* Have severe systemic active infection;
* Have a history of tuberculosis within 1 year before enrollment, or had an active TB infection more than 1 year before but not received adequate anti-TB treatment;
* Human immunodeficiency virus (HIV) positive, syphilis (Anti-TB) positive;
* Known acute or chronic active hepatitis B (HBsAg positive or HBcAb positive, and HBV DNA ≥ 200 IU/mL or ≥ 103 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and positive for HCV RNA test);
* Known impaired gastrointestinal (GI) function or GI diseases that may significantly affect the absorption or metabolism of oral drugs; abdominal fistula, gastrointestinal perforation or abdominal abscess occurred within 6 months before the first administration;
* Subjects taking known moderate or strong inducers and inhibitors of CYP3A within 14 days before the first administration;
* Active autoimmune and inflammatory diseases；
* Women who are pregnant or breastfeeding；
* Subjects who are considered unsuitable for the study judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-02-14 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
Ph Ia/Ib: Overall safety profile including adverse events | Baseline up to approximately 2 years
  * Adverse Events will be graded by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version [5.0])
  * Incidence of Dose Limiting Toxicities
Ph Ia/Ib: Recommended phase 2 doses (RP2D) of XNW29016 | Approximately 12 months
  RP2D of XNW29016 as administered orally twice daily (BID), continuously in 28-day cycles, in subjects by safety data, pharmacokinetic data, pharmacodynamic data and efficacy data

SECONDARY OUTCOMES:
Ph Ia/Ib: Pharmacokinetic Parameters | The cycle 0 and first 28-day cycle of therapy
  The area under the plasma concentration-time curve (AUC)
Ph Ia/Ib: Pharmacokinetic Parameters | The cycle 0 and first 28-day cycle of therapy
  Maximum plasma concentration (Cmax)
Ph Ia/Ib: Pharmacokinetic Parameters | The cycle 0 and first 28-day cycle of therapy
  Elimination half-life (t1/2)
Ph Ia/Ib: Pharmacodynamic Parameters | The cycle 0 and first 28-day cycle of therapy
  The relative change of PAR with the baseline before and after administration
Overall Response Rate (ORR) | Baseline up to approximately 2 years
  ORR was defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR). ORR was based on RECIST 1.1 response for patients with measurable disease at baseline reviewed by the investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- 17 South Li, Panjiayuan, Chaoyang District, Beijing City., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided